CLINICAL TRIAL: NCT04802642
Title: Evaluation of COVID-19 Fear, Anxiety and Their Effects in Physiotherapy Technician Students
Status: Completed | Type: Observational
Sponsor: Ufuk University (Other)
Responsible Party: Principal Investigator, Elzem Bolkan Günaydın, Lecturer Doctor, Ufuk University
Other Study IDs: 2020-4-25
Record Dates: First submitted 2021-03-16; First posted 2021-03-17 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Covid19; Anxiety and Fear
MeSH Terms: conditions — COVID-19; Anxiety Disorders | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey — Survey

SUMMARY:
80 participants studying in the physiotherapy technician department were included in this cross-sectional study. Participants' age, gender, year of being a student, the people they live with, the precautions they take regarding COVID-19, whether there is a history of COVID-19 in them or their immediate surroundings, and whether they have COVID-19 transmission and / or contagion fears during their vocational training, whether there are fears of achieving professional goals and competence because of COVID-19 and / or its consequences were recorded. Afterwards, the participants were asked to answer the questions on the coronavirus anxiety scale, the fear of COVID-19 scale and the cognitive and behavioral avoidance subscales of the Avoidance Attitudes from COVID-19 scale.

ELIGIBILITY:
Inclusion Criteria:

1. Being between the ages of 18-65
2. Being a physiotherapy technician student

Exclusion Criteria:

1. Being under the age of 18, over the age of 65

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 80 volunteers between the ages of 18-65, who are physiotherapy technician students, were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Coronavirus anxiety scale | 2 months
  It is a 5-item scale developed by Lee at all. to evaluate coronavirus-related anxiety. Participants indicate how often they have experienced the situations stated in each item with a 5-point Likert-type scale (0 = none, 1 = rare [less than 1 or 2 days], 2 = several days, 3 = more than 7 days, 4 = last 2 almost everyday a week). The total score is obtained by adding the item scores. The higher total score is higher coronavirus-related anxiety.
The Fear of COVID-19 Scale | 2 months
  It is a 7-item scale developed by Ahorsu et all. to evaluate coronavirus-related fear. Participants indicate how often they experience the situations stated in each item with a 5-point Likert-type scale (1 = strongly disagree, 2 = disagree, 3 = undecided, 4 = agree, 5 = strongly agree). The total score is obtained by summing the item scores, the higher total score is higher the coronavirus-related fear.

CONTACTS AND LOCATIONS:
Overall Officials: elzem Bolkan Günaydın, Principal Investigator — Ufuk University
Locations (1):
- Ufuk University, Ankara, Çankaya, Turkey (Türkiye)